CLINICAL TRIAL: NCT04046809
Title: Effect of Neurotidine® (Citicoline Free Acid in Oral Solution) on Quality of Life in Patients With Glaucoma
Brief Title: Study of Neurotidine® Intake on Life Quality of Patients With Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omikron Italia S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEUQOL2018; 2018-002187-11 (EudraCT Number)
Record Dates: First submitted 2019-07-29; First posted 2019-08-06 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Treatment (Experimental): 500 ml oral solution containing citicoline free acid 50 mg/ml.
  Interventions: Other: Food for special medical purposes: Neurotidine®
- Placebo (Placebo Comparator): 500 ml oral solution indistinguishable from active product in appearance and taste
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Food for special medical purposes: Neurotidine® — Each patient will be given the bottles for the first 3-month treatment period by the hospital pharmacist and will be asked to return them at the end of the period (3 months). Then the patients will be given the other bottles for the next phase of the study (3 months): these will contain placebo if the patient received Neurotidine® in the first phase of the study and vice versa. Again, the patients will be asked to return after 3 months with the study bottles and will be given the last set of bottles for the final phase of the study (3 months).
  Administration at a dosage of 10 ml in the morning.
  Arms: Study Treatment
Other: Placebo — Each patient will be given the bottles for the first 3-month treatment period by the hospital pharmacist and will be asked to return them at the end of the period (3 months). Then the patients will be given the other bottles for the next phase of the study (3 months): these will contain placebo if the patient received Neurotidine® in the first phase of the study and vice versa. Again, the patients will be asked to return after 3 months with the study bottles and will be given the last set of bottles for the final phase of the study (3 months).
  Administration at a dosage of 10 ml in the morning.
  Arms: Placebo

SUMMARY:
The purpose for the study consists in the assessment of the role of Neurotidine® (citicoline oral solution) on the dopaminergic pathway and particularly its potential implications on psychophysical performance and quality of life. Other objectives are the assessment of the tolerability and safety of Neurotidine®.

DETAILED DESCRIPTION:
Primary open angle glaucoma is a chronic progressive neurodegenerative disease and the only proven effective therapy involves reduction of intraocular pressure (IOP). Although treatment effect is quite large, a significant proportion of patients show disease progression with apparently controlled IOP. Given the similarities with other neurodegenerative diseases - particularly in the mechanisms of cell death -neuroprotective treatments have been tried also in glaucoma. Interesting results from experimental studies and weak evidence from human glaucoma trials have been published in recent years. Citicoline is one of the promising molecules with a putative neuroprotective action and has been tried on patients with a number of neurodegenerative diseases with encouraging results. Pilot studies on glaucomatous patients showed a possible effect of citicoline in reducing progression of visual field changes, though these findings need to be confirmed by larger randomized clinical trials.

The aim of this randomized, double-masked, placebo-controlled, cross-over study is to test whether the intake of Neurotidine® (citicoline free acid in oral solution) can be associated with an improvement of quality of life in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be eligible for the study:

* Signed written informed consent.
* Age ≥ 18 years.
* Patients with bilateral open-angle glaucoma (OAG). PEX and pigmentary glaucoma will be included.
* Controlled IOP
* Patients with moderate damage in the better eye, with mean deviation from normal value (MD) ranging from -6 to -12 dB in the 6 months prior to enrollment. At the screening assessment, MD must range from -5 to -13 dB.

Glaucoma definition will be based on visual field (VF) damage (24-2, SITA standard strategy) corresponding to glaucomatous changes at the optic nerve head. Values of IOP will not be an inclusion criterion, though a "controlled IOP" based on the clinician's judgement will be required.

Exclusion Criteria:

Patients must meet none of the following criteria to be eligible for the study:

* Single-eyed patients (visual acuity <0.1 in one eye).
* Patients without the psychophysical requirements to adequately participate and complete the trial.
* Patients with chronic angle-closure glaucoma (CACG) or other types of glaucoma.
* Patients with other ocular comorbidities interfering with the correct assessment of the glaucomatous damage to the VF.
* Patients who have undergone surgery within 6 months.
* Patients taking other potential neuroprotectors, including topical, competing with Neurotidine®.
* Patients with Parkinson's disease, dementia or a diagnosis of stroke in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
The mean change of "intra-patient" global score of the Visual Functioning Questionnaire 25 (VFQ-25) after Neurotidine® vs placebo. | At 6 months compared to baseline
  Primary outcome is based on the global score of the VFQ-25 questionnaire. Specifically, the VFQ-25 consists of a base set of 25 vision targeted questions. The global score derives from the summary of the scores deriving from each question. The total score has a minimum value "0" considered as the worst visual functionality, and the maximum value "100" considered as the better visual functionality.

SECONDARY OUTCOMES:
The change of other scores of the questionnaire: Visual Functioning Questionnaire 25 (VFQ-25). | Up to 9 months compared to baseline
  Other score utilized in the study: general health, general vision, near and far activities, social, mental, role difficulties, etc.
The change of other scores of the questionnaire: Short Form Health Survey - 36 items (SF-36). | Up to 9 months compared to baseline
  Other score utilized in the study: general health, general vision, near and far activities, social, mental, role difficulties, etc.
The safety and tolerability of Neurotidine®. | Up to 9 months compared to baseline
  The safety and tolerability of Neurotidine® will be detected on the basis of possible adverse events. In particular, they will be documented in the CRF. Possible adverse events will be communicated directly by the patient and/or detected by the Investigator during the medical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Rossetti, Prof., Principal Investigator — Presidio Ospedale San Paolo
Locations (5):
- University Hospitals Leuven, Leuven, Belgium
- Aristotle University of Thessaloniki AHEPA Hospital Thessaloniki, Thessaloniki, Greece
- Italy (2):
  - Presidio Ospedale San Paolo, Milan, MI
  - Fondazione PTV Policlinico Tor Vergata, Roma
- CTIG - Teknon, Barcelona, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04046809/Prot_SAP_000.pdf